CLINICAL TRIAL: NCT05582499
Title: Fudan University Shanghai Cancer Center Breast Cancer Precision Platform Series Study- Neoadjuvant Therapy (FASCINATE-N)
Brief Title: Fudan University Shanghai Cancer Center Breast Cancer Precision Platform Series Study- Neoadjuvant Therapy
Acronym: FASCINATE-N
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FASCINATE-N
Record Dates: First submitted 2022-09-25; First posted 2022-10-17 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Breast Neoplasm; Breast Cancer; Breast Tumors; Triple-Negative Breast Cancer (TNBC); HER2-positive Breast Cancer; HER2-negative Breast Cancer; Hormone Receptor Positive Tumor; Hormone Receptor Negative Tumor; Early-stage Breast Cancer; Locally Advanced Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — dalpiciclib; pyrotinib; camrelizumab; pertuzumab; Trastuzumab; Goserelin; Letrozole; Taxes; Carboplatin; Epirubicin; Cyclophosphamide; fluzoparib; apatinib; famitinib; anlotinib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (53):
- L1-1 (Experimental): If patients were hormone receptor-positive (HR+) and HER2-negative (HER2-) defined as similarity network fusion 1(SNF1) subtype
  Interventions: Drug: Dalpiciclib; Drug: Goserelin; Drug: Letrozole
- L1-2 (Active Comparator): If patients were HR+HER2- with SNF1 subtype
  Interventions: Drug: Nab paclitaxel; Drug: Carboplatin
- L2-2 (Active Comparator): If patients were HR+HER2- with SNF2 subtype
  Interventions: Drug: Nab paclitaxel; Drug: Carboplatin
- L3-2 (Active Comparator): If patients were HR+HER2- with SNF3 subtype
  Interventions: Drug: Nab paclitaxel; Drug: Carboplatin
- L4-2 (Active Comparator): If patients were HR+HER2- with SNF4 subtype
  Interventions: Drug: Nab paclitaxel; Drug: Carboplatin
- L4-low-1 (Experimental): If patients were HR+HER2-low with SNF4 subtype
  Interventions: Drug: SHR-A1811
- L4-low-2 (Active Comparator): If patients were HR+HER2-low with SNF4 subtype
  Interventions: Drug: Nab paclitaxel; Drug: Carboplatin
- TN1-1 (Experimental): If patients were triple-negative breast cancer with immunomodulatory (IM) subtype
  Interventions: Drug: Camrelizumab; Drug: Nab paclitaxel; Drug: Carboplatin; Drug: Epirubicin; Drug: Cyclophosphamide
- TN1-2 (Active Comparator): If patients were triple-negative breast cancer with IM subtype
  Interventions: Drug: Nab paclitaxel; Drug: Carboplatin; Drug: Epirubicin; Drug: Cyclophosphamide
- TN2-1 (Experimental): If patients were triple-negative breast cancer with basal-like immune suppressed (BLIS) subtype
  Interventions: Drug: Nab paclitaxel; Drug: Carboplatin; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Fluzoparib
- TN2-2 (Active Comparator): If patients were triple-negative breast cancer with BLIS subtype
  Interventions: Drug: Nab paclitaxel; Drug: Carboplatin; Drug: Epirubicin; Drug: Cyclophosphamide
- TN3-1 (Experimental): If patients were triple-negative breast cancer with androgen receptor positive HER2 activated (AR HER2) subtype
  Interventions: Drug: Pyrotinib; Drug: Nab paclitaxel; Drug: Carboplatin; Drug: Epirubicin; Drug: Cyclophosphamide
- TN3-2 (Active Comparator): If patients were triple-negative breast cancer with AR HER2 subtype
  Interventions: Drug: Nab paclitaxel; Drug: Carboplatin; Drug: Epirubicin; Drug: Cyclophosphamide
- TN4-1.1 (Experimental): If patients were HR-HER2-low
  Interventions: Drug: SHR-A1811
- TN4-2 (Active Comparator): If patients were HR-HER2-low
  Interventions: Drug: Nab paclitaxel; Drug: Carboplatin; Drug: Epirubicin; Drug: Cyclophosphamide
- TN5-1.1 (Experimental): If patients were triple-negative breast cancer with other subtypes
  Interventions: Drug: SHR-A1921
- TN5-2 (Active Comparator): If patients were triple-negative breast cancer with other subtypes
  Interventions: Drug: Nab paclitaxel; Drug: Carboplatin; Drug: Epirubicin; Drug: Cyclophosphamide
- H1-1.1 (Experimental): If patients were HR+HER2+
  Interventions: Drug: Pyrotinib; Drug: SHR-A1811
- H1-2 (Active Comparator): If patients were HR+HER2+
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab; Drug: Nab paclitaxel; Drug: Carboplatin
- H2-1.1 (Experimental): If patients were HR-HER2+
  Interventions: Drug: Pyrotinib
- H2-2 (Active Comparator): If patients were HR-HER2+
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab; Drug: Nab paclitaxel; Drug: Carboplatin
- L2-1.2 (Experimental): If patients were HR+HER2- with similarity network fusion 2 (SNF2) subtype
  Interventions: Drug: SHR-1316; Drug: Nab paclitaxel; Drug: Carboplatin
- L3-1.2 (Experimental): If patients were HR+HER2- with similarity network fusion 3 (SNF3) subtype
  Interventions: Drug: Nab paclitaxel; Drug: Carboplatin; Drug: Fluzoparib
- L4-1.2 (Experimental): If patients were HR+HER2- with similarity network fusion 4 (SNF4) subtype
  Interventions: Drug: Nab paclitaxel; Drug: Carboplatin; Drug: Apatinib
- TN5-1.2 (Experimental): If patients were triple-negative breast cancer with other subtypes
  Interventions: Drug: SHR-1316; Drug: SHR-A1921
- H1-1.2 (Experimental): If patients were HR+HER2+
  Interventions: Drug: SHR-A1811
- H2-1.2 (Experimental): If patients were HR-HER2+
  Interventions: Drug: Pyrotinib; Drug: SHR-A1811
- TN4-1.2 (Experimental): If patients were HR-HER2-low
  Interventions: Drug: SHR-A1811; Drug: Camrelizumab; Drug: Famitinib
- L2-1.1 (Experimental): If patients were HR+HER2- with similarity network fusion 2 (SNF2) subtype
  Interventions: Drug: Dalpiciclib; Drug: Goserelin; Drug: Letrozole
- L2-1.3 (Experimental): If patients were HR+HER2- with similarity network fusion 2 (SNF2) subtype
  Interventions: Drug: SHR-1316; Drug: Nab paclitaxel; Drug: Carboplatin; Drug: Famitinib
- L3-1.1 (Experimental): If patients were HR+HER2- with similarity network fusion 3 (SNF3) subtype
  Interventions: Drug: Dalpiciclib; Drug: Goserelin; Drug: Letrozole
- L4-1.1 (Experimental): If patients were HR+HER2- with similarity network fusion 4 (SNF4) subtype
  Interventions: Drug: SHR-A1921
- L5-1 (Experimental): If patients were HR+HER2-
  Interventions: Drug: Cyclophosphamide; Drug: HB1801; Drug: LEM
- L5-2 (Experimental): If patients were HR+HER2-
  Interventions: Drug: Cyclophosphamide; Drug: HB1801; Drug: LEM
- L6 (Experimental): If patients were HR+HER2-low
  Interventions: Drug: SHR-A1811; Drug: SHR-1316; Drug: Famitinib
- L7 (Experimental): If patients were HR+HER2-low
  Interventions: Drug: Famitinib; Drug: TQB2102; Drug: Benmelstobart
- L8 (Experimental): If patients were HR+HER2-
  Interventions: Drug: TQB2102; Drug: Anlotinib; Drug: TQB2868
- L9 (Experimental): If patients were HR+HER2-low
  Interventions: Drug: Nab paclitaxel; Drug: Carboplatin; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Ivonescimab
- TN6-1 (Experimental): TNBC
  Interventions: Drug: SHR-A1811; Drug: SHR-1316; Drug: Famitinib
- TN6-2 (Experimental): TNBC
  Interventions: Drug: SHR-A1811; Drug: SHR-1316
- TN7-1 (Experimental): If patients were HR-HER2-low
  Interventions: Drug: TQB2102; Drug: Benmelstobart
- TN7-2 (Experimental): If patients were HR-HER2-low
  Interventions: Drug: TQB2102; Drug: Benmelstobart; Drug: Anlotinib
- TN8 (Experimental): TNBC
  Interventions: Drug: TQB2102; Drug: TQB2868
- TN9 (Experimental): TNBC
  Interventions: Drug: Carboplatin; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: paclitaxel
- H3 (Experimental): If patients were HER2+
  Interventions: Drug: JSKN003
- H4-1 (Experimental): If patients were HER2+
  Interventions: Drug: SHR-A1811; Drug: Pertuzumab; Drug: Trastuzumab; Drug: Nab paclitaxel; Drug: Carboplatin
- H4-2 (Experimental): If patients were HER2+
  Interventions: Drug: SHR-A1811
- H4-3 (Experimental): If patients were HER2+
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab; Drug: Nab paclitaxel; Drug: Carboplatin
- H4-4 (Experimental): If patients were HER2+
  Interventions: Drug: Pyrotinib; Drug: SHR-A1811
- H5 (Experimental): If patients were HER2+
  Interventions: Drug: SHR-A1811; Drug: SHR-4602
- H6-1 (Experimental): If patients were HER2+
  Interventions: Drug: SHR-A1811; Drug: HRS-4508
- H6-2 (Experimental): If patients were HER2+
  Interventions: Drug: SHR-A1811; Drug: Pertuzumab; Drug: HRS-4508
- L10 (Experimental): If patients were HR+HER2-
  Interventions: Drug: Nab paclitaxel; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: JS207

INTERVENTIONS:
Drug: Dalpiciclib — an oral cyclin-dependent kinases (CDK) 4/6 inhibitor
  Other Names: SHR-6390
  Arms: L1-1; L2-1.1; L3-1.1
Drug: Pyrotinib — an irreversible dual pan-erbb receptor tyrosine kinase receptor tyrosine kinase (ERBB) inhibitor
  Arms: H1-1.1; H2-1.1; H2-1.2; H4-4; TN3-1
Drug: SHR-A1811 — an anti-HER2 antibody-drug conjugate (ADC)
  Arms: H1-1.1; H1-1.2; H2-1.2; H4-1; H4-2; H4-4; H5; H6-1; H6-2; L4-low-1; L6; TN4-1.1; TN4-1.2; TN6-1; TN6-2
Drug: SHR-1316 — an anti-programmed death ligand 1 (PD-L1) antibody
  Arms: L2-1.2; L2-1.3; L6; TN5-1.2; TN6-1; TN6-2
Drug: Camrelizumab — an anti-programmed death-1 (PD1) antibody
  Other Names: SHR-1210
  Arms: TN1-1; TN4-1.2
Drug: SHR-A1921 — Trophoblast cell-surface antigen 2 (TROP2) ADC
  Arms: L4-1.1; TN5-1.1; TN5-1.2
Drug: Pertuzumab — Pertuzumab
  Arms: H1-2; H2-2; H4-1; H4-3; H6-2
Drug: Trastuzumab — Trastuzumab
  Arms: H1-2; H2-2; H4-1; H4-3
Drug: Goserelin — goserelin
  Arms: L1-1; L2-1.1; L3-1.1
Drug: Letrozole — letrozole
  Arms: L1-1; L2-1.1; L3-1.1
Drug: Nab paclitaxel — Albumin paclitaxel
  Arms: H1-2; H2-2; H4-1; H4-3; L1-2; L10; L2-1.2; L2-1.3; L2-2; L3-1.2; L3-2; L4-1.2; L4-2; L4-low-2; L9; TN1-1; TN1-2; TN2-1; TN2-2; TN3-1; TN3-2; TN4-2; TN5-2
Drug: Carboplatin — Carboplatin
  Arms: H1-2; H2-2; H4-1; H4-3; L1-2; L2-1.2; L2-1.3; L2-2; L3-1.2; L3-2; L4-1.2; L4-2; L4-low-2; L9; TN1-1; TN1-2; TN2-1; TN2-2; TN3-1; TN3-2; TN4-2; TN5-2; TN9
Drug: Epirubicin — Epirubicin
  Arms: L10; L9; TN1-1; TN1-2; TN2-1; TN2-2; TN3-1; TN3-2; TN4-2; TN5-2; TN9
Drug: Cyclophosphamide — Cyclophosphamide
  Arms: L10; L5-1; L5-2; L9; TN1-1; TN1-2; TN2-1; TN2-2; TN3-1; TN3-2; TN4-2; TN5-2; TN9
Drug: Fluzoparib — an original poly adenosine diphosphate-ribose polymerase (PARP) inhibitor
  Other Names: SHR-3162
  Arms: L3-1.2; TN2-1
Drug: Apatinib — tyrosine kinase inhibitors
  Arms: L4-1.2
Drug: Famitinib — tyrosine kinase inhibitors
  Arms: L2-1.3; L6; L7; TN4-1.2; TN6-1
Drug: HB1801 — Albumin docetaxel
  Arms: L5-1; L5-2
Drug: LEM — liposome-entrapped mitoxantrone
  Arms: L5-1; L5-2
Drug: TQB2102 — an anti-HER2 ADC
  Arms: L7; L8; TN7-1; TN7-2; TN8
Drug: Benmelstobart — an anti-PDL1 antibody
  Arms: L7; TN7-1; TN7-2
Drug: Anlotinib — an tyrosine kinase inhibitor
  Arms: L8; TN7-2
Drug: TQB2868 — anti-PD-1/TGF-βRII
  Arms: L8; TN8
Drug: Ivonescimab — an anti-PD-1/VEGF bispecific antibody
  Arms: L9
Drug: JS207 — an anti-PD-1/VEGF bispecific antibody
  Arms: L10
Drug: JSKN003 — an anti-HER2 ADC
  Arms: H3
Drug: HRS-4508 — an HER2 inhibitor
  Arms: H6-1; H6-2
Drug: SHR-4602 — an anti-HER2 ADC
  Arms: H5
Drug: paclitaxel — paclitaxel
  Arms: TN9

SUMMARY:
The purpose of this study is to establish a prospective, single-center platform research based on clinical subtypes to explore precision neoadjuvant therapy in patients with operable breast cancer who met the indications for neoadjuvant chemotherapy and by the update of basic translational research in the center, especially the refinement of typing, the discovery of new targets and the development of novel targeted drugs, verified the effectiveness of new targeted drugs in neoadjuvant therapy.

DETAILED DESCRIPTION:
FASCINATE-N is a platform that will compare the efficacy of novel drugs alone or in combination with standard chemotherapy with the efficacy of standard therapy alone. The goal is to identify improved treatment regimens for subsets on the basis of clinical subtyping. In this trial, breast cancer patients eligible for inclusion can be randomly divided into the precision treatment group and conventional neoadjuvant chemotherapy group according to molecular typing and subtyping. The research therapy arm can be updated with the update of basic translational research in our center, especially the refinement of typing, the discovery of new targets and the development of novel targeted drugs. As described for previous adaptive trials, regimens that show to be more effective than standard therapy will graduate from the trial with their corresponding biomarker signature(s). Regimens will be dropped if they show a low probability of improved efficacy with any biomarker signature. New drugs will enter as those that have undergone testing complete their evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive cancer of the breast and meet the clinical stage II（T2N0-1M0/T3N0M0）or III（T2N2M0/T3N1-2M0) criteria;
* Age between18-70 years;
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
* ER, PR and HER2 status were measured by immunohistochemistry (IHC);
* LVEF≥55%；
* Definition of SNF subtypes: SNF subtypes confirmed by digital pathology of H&E slices;
* Triple negative subtyping: On the basis of triple-negative pathological diagnosis, AR, cluster of differentiation 8 (CD8) and Forkhead Box C1 (FOXC1) were combined to define the subtyping;
* At least one measurable lesion according to RECIST version 1.1
* Normal organ and marrow function: Hemoglobin (HB) ≥90 g/L (No blood was transfused within 14 days), Absolute neutrophil count ≥ 1500/μL, Platelets ≥ 75,000/μL, Total bilirubin ≤ 1.5 x ULN), aspartate aminotransferase (AST) (SGOT) and alanine aminotransferase (ALT) (SGPT) ≤ 3 x ULN, creatinine < 1 x ULN, endogenous creatinine clearance > 50 ml/min (Cockcroft-Gault formula);
* Non-pregnant and non-lactating, fertile female subjects were required to use a medically approved contraceptive method for the duration of the study treatment and at least 3 months after the last use of the study drug;
* Ability to understand and willingness to sign a written informed consent

Exclusion Criteria:

* Previous cytotoxic chemotherapy, endocrine therapy, biological therapy or radiotherapy for any reason;
* Patients with New York Heart Association (NYHA) grade II or above heart disease (including grade II);
* Patients with severe systemic infections or other serious diseases;
* Patients with known allergy or intolerance to the study drug or its excipients;
* Other malignant tumors in the past 5 years, except cured cervical carcinoma in situ and non-melanoma skin cancer;
* Pregnant or lactating patients of childbearing age who refused to take appropriate contraceptive measures during the course of the study;
* Participated in other trial studies within 30 days before the administration of the first dose of the study drug;
* Patients who were judged by the investigator to be unsuitable for this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 716 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR) | through study completion, up to 24 weeks
  Pathological complete response rate

SECONDARY OUTCOMES:
invasive disease-free survival (iDFS) | Three-year Post-surgery Follow-up
  To determine three-year invasive disease-free survival (iDFS) among the treatment arms
Overall response rate (ORR) | up to 24 weeks
  Complete response (CR) + partial response (PR)
CTCAE scale (V4.0) | through study completion, an average of 1 year
  4) To evaluate the rate of adverse effects of patient by the standard CTCAE scale (V4.0)
Evaluate gene expression profile during treatment | through study completion, up to 24 weeks
  To measure gene expression profile of baseline and sequential tumor samples during treatment, through RNA-seq platform
Number of peripheral blood mononuclear cells (PBMC) count during treatment | through study completion, up to 24 weeks
  To measure number of peripheral blood mononuclear cells (PBMC) count from baseline and sequential blood samples during treatment, through Flow CytoMetry platform

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, Professor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center Shanghai, China, 200032, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zuo WJ, Chen L, Shen Y, Wang ZH, Liu GY, Yu KD, Di GH, Wu J, Li JJ, Shao ZM. Rational and trial design of FASCINATE-N: a prospective, randomized, precision-based umbrella trial. Ther Adv Med Oncol. 2024 Feb 14;16:17588359231225032. doi: 10.1177/17588359231225032. eCollection 2024. PMID 38362377